CLINICAL TRIAL: NCT03463863
Title: The Safety And Efficacy Of Autologus Rectus Sheath Fascia As A Midurethral Transobturator Tension Free Vaginal Tape For Treatment Of Stress Urinary Incontinence.
Brief Title: Midurethral Sling With Autologus Rectus Sheath
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: sarah mohamed hassan (Other)
Responsible Party: Sponsor-Investigator, sarah mohamed hassan, lecturer of obstetrics and gynecology, Kasr El Aini Hospital
Organization: Kasr El Aini Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 732222
Record Dates: First submitted 2018-03-07; First posted 2018-03-13 (Actual); Last update posted 2018-03-16 (Actual); Status verified 2018-03

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: rectus sheath midurethral sling

SUMMARY:
assessment of the safety and efficacy surgeon tailored rectus sheath midurethral sling

DETAILED DESCRIPTION:
the rectus sheath is harvested in 5 cm length and 2 cm width , A 2cm width 8 cm length polypropolyine mesh is attached to the harvest rectus sheet sling on both side The procedure is carried with a similar technique to the outside in TOT.

ELIGIBILITY:
Inclusion Criteria:

* stress incontinence

Exclusion Criteria:

* overactive bladder

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-08-10 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
cure rate of stress incontinence | one year after surgery
  history and urodynamic study

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr El Ainiy Hospital, Cairo, Egypt